CLINICAL TRIAL: NCT01217229
Title: A Phase 2 Safety and Efficacy Study of Orally Administered PLX3397 in Adults With Relapsed or Refractory Hodgkin Lymphoma
Brief Title: Safety and Efficacy Study of PLX3397 in Adults With Relapsed or Refractory Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Plexxikon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLX108-03
Record Dates: First submitted 2010-10-04; First posted 2010-10-08 (Estimated); Results first posted 2013-03-15 (Estimated); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Hodgkin Lymphoma
Keywords: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — pexidartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PLX3397 (Experimental)
  Interventions: Drug: PLX3397

INTERVENTIONS:
Drug: PLX3397 — Capsules administered once or twice daily, continuous dosing. Subjects will begin with 900 mg/day, but should safety data allow in our PLX108-01 study, subject may dose at 1200 mg/day.

SUMMARY:
PLX3397 is a selective inhibitor of Fms, Kit, and oncogenic Flt3 activity.The primary objective of this study is to evaluate the efficacy, as measured by overall response rate, of orally administered PLX3397 in patients with relapsed or refractory classical Hodgkin lymphoma (HL). Secondary objectives include safety, the duration of response, the disease control rate, progression free survival, and how the drug affects your body.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥18 years old
2. Pathologic confirmation of relapsed or refractory classical Hodgkin lymphoma, with archival or fresh tissue available for retrospective analysis.
3. Patients must have progressed after-or been ineligible for-autologous stem cell transplantation. Patients who received a prior allogeneic stem cell transplantation are eligible if they have no evidence of graft versus host disease (GVHD) and have been off immunosuppression for at least 3 months prior to Cycle 1 Day 1 (C1D1).
4. Documented disease that is radiographically measurable (≥2 cm in the largest transverse dimension).
5. Patients must have discontinued any previous monoclonal antibody, radioimmunotherapy, or cytotoxic chemotherapy at least 28 days prior to C1D1 and must have recovered fully from the side effects of that treatment prior to beginning study treatment.
6. Women of child-bearing potential must have a negative pregnancy test within 7 days of initiation of dosing and must agree to use an acceptable method of birth control while on study drug and for 3 months after the last dose. Women of non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥1 year. Men of child-bearing potential must also agree to use an acceptable method of birth control while on study drug.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
8. Adequate hematologic, hepatic, and renal function (absolute neutrophil count ≥1.0 x 109/L, Hgb >9 g/dL, platelet count ≥50 x 109/L, Aspartate Transaminase (AST) / Alanine Transaminase (ALT) ≤2.5x Upper limit of normal (ULN), creatinine ≤1.5x ULN)
9. Willing and able to provide written informed consent prior to any study related procedures and to comply with all study requirements

Exclusion Criteria:

1. Investigational drug use within 28 days of the first dose of PLX3397
2. History or clinical evidence of central nervous system, meningeal, or epidural disease including brain metastasis
3. Patients with another active cancer [excluding basal cell carcinoma or cervical intraepithelial neoplasia (cervical carcinoma in situ) or melanoma in situ]. Prior history of other cancer is allowed, as long as there was no active disease within the prior 5 years.
4. Patients with uncontrolled intercurrent illness, an active or uncontrolled infection, or a fever >38.5˚C (not due to tumor fever) on C1D1
5. Refractory nausea and vomiting, malabsorption, biliary shunt, or significant bowel resection that would preclude adequate absorption
6. Patients with serious illnesses, medical conditions, or other medical history including abnormal laboratory results, which in the investigator's opinion would be likely to interfere with a patient's participation in the study, or with the interpretation of the results
7. Women of child-bearing potential who are pregnant or breast feeding
8. Corrected QT interval (QTc) ≥450 msec.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-03-03 (Actual); Primary Completion 2012-04-26 (Actual); Study Completion 2012-04-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - UCLA Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Northwestern University, The Robert H Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 20 participants who met all inclusion and no exclusion criteria were enrolled and received treatment at 6 clinic sites in the United States.
Groups:
- PLX3397: Participants received PLX3397 administered once or twice daily with continuous dosing at 900 mg/day.
Period: Overall Study
Arm/Group | PLX3397
Started | 20
Completed | 0
Not Completed | 20
Not completed — Adverse Event | 1
Not completed — Disease progression, deterioration | 2
Not completed — Disease progression, Cheson criteria | 14
Not completed — Protocol Violation | 1
Not completed — Disease progression not confirmed | 2

BASELINE CHARACTERISTICS:
Arm/Group | PLX3397
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (19.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival According to the Cheson Criteria by Kaplan-Meier Analysis Following Orally Administered PLX3397 in Adults With Relapsed or Refractory Hodgkin Lymphoma (Modified Intent-to-Treat Population)
Description: Progression-free survival was assessed by Kaplan Meier analysis and was defined as the number of days from the first day of treatment to the date of first documented disease progression or date of death (whichever occurred first).
Time Frame: Baseline to 1 year postdose
Population: Progression-free survival was assessed in the Modified Intent-to-Treat population.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | PLX3397
Number analyzed (Participants) | 20
days | 56 [54 to 57]

2. Primary Outcome: Summary of Overall Tumor Response and By Cycle Following Orally Administered PLX3397 in Adults With Relapsed or Refractory Hodgkin Lymphoma (Modified Intent-to-Treat Population)
Description: Subjects were monitored for response and disease progression with contrast Computed tomography (CT) /18Fluorodeoxyglucose (FDG)-positron emission tomography (PET) scans every two cycles. Each cycle is 28 days. Response to treatment as defined by Cheson criteria was reported via descriptive statistics. Target tumor response is Complete Response (CR) + Partial Response (PR) and target tumor disease control rate (CR + PR + Stable Disease (SD)) are reported. Per Cheson Criteria, CR is disappearance of all evidence of disease; Partial Response is regression of measurable disease and no new sites (≥50% decrease in sum of product diameters of up to 6 largest dominant masses and splenic/liver nodules), and no increase in size of other nodes/liver/spleen; reduction in target lesions, no growth of non-target or new lesions; Progression is any new lesion or increase by ≥50% of previously involved sites from the nadir.
Time Frame: Baseline to Cycles 3, 5, 7, 10, and 13, up to 1 year postdose
Population: Tumor response was assessed in the Modified Intent-to-Treat population.
Measure: Count of Participants; unit: Participants
Arm/Group | PLX3397
Number analyzed (Participants) | 20
Participants
  Overall: Target tumor response (CR+PR) | 1
  Overall: Target tumor DCR (CR+PR+SD) | 4
  Overall: Complete response (CR) | 0
  Overall: Partial response (PR) | 1
  Overall: Stable disease (SD) | 3
  Overall: Relapsed disease or progressive disease | 13
  Cycle 3: Target tumor response (CR+PR) | 0
  Cycle 3: Target tumor DCR (CR+PR+SD) | 4
  Cycle 3: Complete response (CR) | 0
  Cycle 3: Partial response (PR) | 0
  Cycle 3: Stable disease (SD) | 4
  Cycle 3: Relapsed disease or progressive disease | 1
  Cycle 5: Target tumor response (CR+PR) | 0
  Cycle 5: Target tumor DCR (CR+PR+SD) | 1
  Cycle 5: Complete response (CR) | 0
  Cycle 5: Partial response (PR) | 0
  Cycle 5: Stable disease (SD) | 1
  Cycle 5: Relapsed disease or progressive disease | 0
  Cycle 7: Target tumor response (CR+PR) | 1
  Cycle 7: Target tumor DCR (CR+PR+SD) | 1
  Cycle 7: Complete response (CR) | 0
  Cycle 7: Partial response (PR) | 1
  Cycle 7: Stable disease (SD) | 0
  Cycle 7: Relapsed disease or progressive disease | 0
  Cycle 10: Target tumor response (CR+PR) | 1
  Cycle 10: Target tumor DCR (CR+PR+SD) | 1
  Cycle 10: Complete response (CR) | 0
  Cycle 10: Partial response (PR) | 1
  Cycle 10: Stable disease (SD) | 0
  Cycle 10: Relapsed disease or progressive disease | 0
  Cycle 13: Target tumor response (CR+PR) | 1
  Cycle 13: Target tumor DCR (CR+PR+SD) | 1
  Cycle 13: Complete response (CR) | 0
  Cycle 13: Partial response (PR) | 1
  Cycle 13: Stable disease (SD) | 0
  Cycle 13: Relapsed disease or progressive disease | 0

3. Primary Outcome: Participants With Treatment-Emergent Adverse Events Occurring at a Frequency of ≥10% in Any Preferred Term (Safety Population)
Time Frame: Baseline to 1 year post-dose
Population: Adverse events were assessed in the Safety Analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | PLX3397
Number analyzed (Participants) | 20
Participants
  At least 1 adverse event | 20
  Anaemia | 6
  Thrombocytopenia | 6
  Diarrhoea | 2
  Nausea | 2
  Vomiting | 2
  Chills | 2
  Fatigue | 8
  Pyrexia | 4
  Aspartate aminotransferase increased | 2
  Blood lactate dehydrogenase increased | 5
  Decreased appetite | 3
  Back pain | 2
  Dizziness | 2
  Headache | 2
  Cough | 3
  Dyspnoea | 5
  Productive cough | 2
  Hair colour changes | 8
  Rash | 5

4. Primary Outcome: Participants With at Least Grade 2 Severity Adverse Events by Preferred Term (Safety Population)
Description: Grade 2 adverse events were defined as events that were moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL).
Time Frame: Baseline to 1 year postdose
Population: Adverse events were assessed in the Safety Analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | PLX3397
Number analyzed (Participants) | 20
Participants
  At least 1 Grade 2 adverse event | 13
  At least 1 Grade 3 adverse event | 5
  Grade 2 Anaemia | 6
  Grade 2 Neutropenia | 1
  Grade 3 Neutropenia | 1
  Grade 2 Thrombocytopenia | 1
  Grade 3 Thrombocytopenia | 1
  Grade 2 Fatigue | 5
  Grade 2 Pyrexia | 2
  Grade 3 Lung infection | 1
  Grade 2 Pneumonia | 1
  Grade 3 Blood alkaline phosphatase | 1
  Grade 2 Blood lactate dehydrogenase increased | 2
  Grade 3 Neutrophil count decreased | 3
  Grade 2 Decreased appetite | 1
  Grade 2 Muscular weakness | 1
  Grade 2 Squamous cell carcinoma | 1
  Grade 3 Syncope | 1
  Grade 2 Anxiety | 1
  Grade 2 Dyspnoea | 2
  Grade 2 Erythema multiforme | 1
  Grade 2 Rash | 2
  Grade 3 Rash | 1
  Grade 2 Skin exfoliation | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from study enrollment up to 1 year post dose.
Arm/Group | PLX3397
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PLX3397 (N=20)
Lung infection (Infections and infestations) | 1
Pyrexia (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PLX3397 (N=20)
Anaemia (Blood and lymphatic system disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Fatigue (General disorders) | 8
Hair depigmentation (Skin and subcutaneous tissue disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Eye swelling (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Asthenia (Gastrointestinal disorders) | 1
Chills (Gastrointestinal disorders) | 2
Face odema (Gastrointestinal disorders) | 1
Fatigue (Gastrointestinal disorders) | 8
Pyrexia (Gastrointestinal disorders) | 4
Clostridial infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Blood alkaline phosphatase (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 5
Neutrophil count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Balance disorder (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Menstruation irregular (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Hair colour changes (Skin and subcutaneous tissue disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days